CLINICAL TRIAL: NCT03294850
Title: Evaluation of Biomarkers to Quantify Liver Pathology in Patients With Presumed Non-Alcoholic Steatohepatitis at Baseline and Following Bariatric Surgery (BARI)
Brief Title: Biomarkers of Liver Pathology in Patients With Presumed Non-Alcoholic Steatohepatitis Following Bariatric Surgery
Acronym: BARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMDFH 1000376
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; NAFLD - Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NASH group (Experimental): These are individuals that have been identified as having NASH by MRE. Confirmation with liver biopsy required for continuation in the longitudinal study.
  Interventions: Procedure: Bariatric surgery; Device: HepQuant SHUNT Dual Cholate Liver Diagnostic Kit
- Non-NASH (NAFLD or normal) group (Active Comparator): These are individuals that do not have NASH. They either have normal liver physiology or only have evidence of hepatic steatosis. This group will be studied up until the day of their bariatric surgery and will serve as a comparator population with respect to baseline measurements.
  Interventions: Procedure: Bariatric surgery; Device: HepQuant SHUNT Dual Cholate Liver Diagnostic Kit

INTERVENTIONS:
Procedure: Bariatric surgery — Subjects enrolling in the study who are undergoing bariatric surgery as part of their medical care will be studied
Device: HepQuant SHUNT Dual Cholate Liver Diagnostic Kit — For the experimental group, the device will be used to monitor the effect of bariatric surgery on liver function. For the active comparator group, the device will be used for the assessment of baseline liver function.

SUMMARY:
The purpose of this study is to evaluate imaging and other biomarkers of non-alcoholic fatty liver disease before and after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Undergoing bariatric surgery (Roux-en-Y or gastric sleeve only) as part of clinical care.
* Negative human chorionic gonadotropin (hCG) level (female participants who become pregnant during the study will be withdrawn)
* For nonalcoholic steatohepatitis (NASH) participants - FibroScan: Controlled Attenuation Parameter (CAP) 290 db/m and Vibration-Controlled Transient Elastography (VCTE) 8 kilopascal (kPa). For participants who meet FibroScan criteria, inclusion will require MRI-PDFF ≥8%; MRE: ≥2.7 kPa.
* For NAFLD or normal participants - FibroScan: No requirement for minimum CAP level and VCTE <7 kPa. For participants that meet the FibroScan criteria- no requirement for minimum MRI-PDFF; MRE ≤ 2 kPa.
* Histopathology assessment of liver biopsy that confirms NASH diagnosis
* Hemoglobin A1c (HbA1c) ≤ 9.5%
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L)
* Body mass index (BMI) ≥ 35 kg/m2
* Able to speak and understand written and spoken English
* Understands the procedures and agrees to participate by giving written informed consent
* Willing and able to comply with scheduled visits, laboratory tests, and other study procedures

Exclusion Criteria:

* Participation in other studies involving investigational drug(s) within 30 days prior to Screening Visit 1
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males within the previous 6 months
* A total score of 8 on the Alcohol Use Disorders Identification Test questionnaire (Appendix B), indicating harmful or hazardous ethanol consumption
* A positive urine drug test for illicit drugs
* Clinical evidence of hepatic decompensation, including, but not limited to esophageal varices, ascites, or hepatic encephalopathy
* Evidence of other forms of chronic liver disease (including laboratory tests as assessed by a sponsor-identified laboratory, and confirmed with a single repeat, if needed): Hepatitis B virus (HBV): defined by presence of hepatitis B surface antigen (HBsAg); Hepatitis C virus (HCV): As defined by a clinical history of previous diagnosis of Hepatitis C (treated or untreated) or a positive Hepatitis C antibody (HCVAb); Known diagnosis of primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis, or overlap syndrome; Alcoholic liver disease; Known diagnosis of hemochromatosis; Prior known drug-induced liver injury; Known or suspected hepatocellular carcinoma (HCC) or other liver cancer; History of liver transplant, current placement on a liver transplant list, or current model of end-stage liver disease (MELD) score >12; Histological presence of cirrhosis on a prior biopsy.
* Human Immunodeficiency Virus (HIV) infection, defined as presence of HIV antibody
* Diagnosis of type 1 diabetes mellitus
* Any malignancy not considered cured, except basal cell carcinoma and squamous cell carcinoma of the skin (a subject is considered cured if there has been no evidence of cancer recurrence in the previous 5 years)
* Use of drugs historically associated with non-alcoholic fatty liver disease (NAFLD) for 1 month in the previous year prior to Visit 3 (day of Surgery); examples include: amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, other known hepatotoxins
* Subjects with history of severe claustrophobia impacting ability to perform MRI during the study without mild sedation/treatment with an anxiolytic
* Subjects who fulfill any of the contraindications for MRI; examples include metal implants, devices, paramagnetic objects contained within the body and excessive or metal-containing tattoos
* Unable to participate in MR assessments due to physical limitations of equipment tolerances (MRI bore size and 500-pound weight limit) based on Investigator's judgment at screening
* Any person unable to lie still within the environment of the MRI scanner or maintain a breath hold for the required period to acquire images without mild sedation/treatment with an anxiolytic
* Subjects with any anatomical or pathological abnormality that would either preclude or tend to confound the analysis of study data, including any clinically significant abnormal findings on the MRI obtained at Screening Visit 2.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to Screening Visit 1 (participants may not donate blood any time during the study, through the final study visit)
* Known history or suspected hypersensitivity to human serum albumin, or its preparations.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Smith, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed MH, Abu EO, Byrne CD. Non-Alcoholic Fatty Liver Disease (NAFLD): new challenge for general practitioners and important burden for health authorities? Prim Care Diabetes. 2010 Oct;4(3):129-37. doi: 10.1016/j.pcd.2010.02.004. Epub 2010 Mar 17. PMID 20299294
- [Background] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Sanyal AJ, Friedman SL, McCullough AJ, Dimick-Santos L; American Association for the Study of Liver Diseases; United States Food and Drug Administration. Challenges and opportunities in drug and biomarker development for nonalcoholic steatohepatitis: findings and recommendations from an American Association for the Study of Liver Diseases-U.S. Food and Drug Administration Joint Workshop. Hepatology. 2015 Apr;61(4):1392-405. doi: 10.1002/hep.27678. Epub 2015 Mar 19. PMID 25557690
- [Background] Cohen JC, Horton JD, Hobbs HH. Human fatty liver disease: old questions and new insights. Science. 2011 Jun 24;332(6037):1519-23. doi: 10.1126/science.1204265. PMID 21700865
- [Background] Ratziu V, Charlotte F, Heurtier A, Gombert S, Giral P, Bruckert E, Grimaldi A, Capron F, Poynard T; LIDO Study Group. Sampling variability of liver biopsy in nonalcoholic fatty liver disease. Gastroenterology. 2005 Jun;128(7):1898-906. doi: 10.1053/j.gastro.2005.03.084. PMID 15940625
- [Background] Alkhouri N, McCullough AJ. Noninvasive Diagnosis of NASH and Liver Fibrosis Within the Spectrum of NAFLD. Gastroenterol Hepatol (N Y). 2012 Oct;8(10):661-8. PMID 24683373
- [Background] Papagianni M, Sofogianni A, Tziomalos K. Non-invasive methods for the diagnosis of nonalcoholic fatty liver disease. World J Hepatol. 2015 Apr 8;7(4):638-48. doi: 10.4254/wjh.v7.i4.638. PMID 25866601
- [Background] Dulai PS, Sirlin CB, Loomba R. MRI and MRE for non-invasive quantitative assessment of hepatic steatosis and fibrosis in NAFLD and NASH: Clinical trials to clinical practice. J Hepatol. 2016 Nov;65(5):1006-1016. doi: 10.1016/j.jhep.2016.06.005. Epub 2016 Jun 14. PMID 27312947
- [Background] Hashemi SA, Alavian SM, Gholami-Fesharaki M. Assessment of transient elastography (FibroScan) for diagnosis of fibrosis in non-alcoholic fatty liver disease: A systematic review and meta-analysis. Caspian J Intern Med. 2016 Fall;7(4):242-252. PMID 27999641
- [Background] Barker KB, Palekar NA, Bowers SP, Goldberg JE, Pulcini JP, Harrison SA. Non-alcoholic steatohepatitis: effect of Roux-en-Y gastric bypass surgery. Am J Gastroenterol. 2006 Feb;101(2):368-73. doi: 10.1111/j.1572-0241.2006.00419.x. PMID 16454845
- [Background] Rabl C, Campos GM. The impact of bariatric surgery on nonalcoholic steatohepatitis. Semin Liver Dis. 2012 Feb;32(1):80-91. doi: 10.1055/s-0032-1306428. Epub 2012 Mar 13. PMID 22418890
- [Background] Hafeez S, Ahmed MH. Bariatric surgery as potential treatment for nonalcoholic fatty liver disease: a future treatment by choice or by chance? J Obes. 2013;2013:839275. doi: 10.1155/2013/839275. Epub 2013 Jan 29. PMID 23431426
- [Background] Schneck AS, Anty R, Patouraux S, Bonnafous S, Rousseau D, Lebeaupin C, Bailly-Maitre B, Sans A, Tran A, Gugenheim J, Iannelli A, Gual P. Roux-En Y Gastric Bypass Results in Long-Term Remission of Hepatocyte Apoptosis and Hepatic Histological Features of Non-alcoholic Steatohepatitis. Front Physiol. 2016 Aug 19;7:344. doi: 10.3389/fphys.2016.00344. eCollection 2016. PMID 27594839
- [Background] Alizai PH, Wendl J, Roeth AA, Klink CD, Luedde T, Steinhoff I, Neumann UP, Schmeding M, Ulmer F. Functional Liver Recovery After Bariatric Surgery--a Prospective Cohort Study with the LiMAx Test. Obes Surg. 2015 Nov;25(11):2047-53. doi: 10.1007/s11695-015-1664-0. PMID 25869925
- [Background] Barr J, Caballeria J, Martinez-Arranz I, Dominguez-Diez A, Alonso C, Muntane J, Perez-Cormenzana M, Garcia-Monzon C, Mayo R, Martin-Duce A, Romero-Gomez M, Lo Iacono O, Tordjman J, Andrade RJ, Perez-Carreras M, Le Marchand-Brustel Y, Tran A, Fernandez-Escalante C, Arevalo E, Garcia-Unzueta M, Clement K, Crespo J, Gual P, Gomez-Fleitas M, Martinez-Chantar ML, Castro A, Lu SC, Vazquez-Chantada M, Mato JM. Obesity-dependent metabolic signatures associated with nonalcoholic fatty liver disease progression. J Proteome Res. 2012 Apr 6;11(4):2521-32. doi: 10.1021/pr201223p. Epub 2012 Mar 15. PMID 22364559
- [Background] Nielsen MJ, Nedergaard AF, Sun S, Veidal SS, Larsen L, Zheng Q, Suetta C, Henriksen K, Christiansen C, Karsdal MA, Leeming DJ. The neo-epitope specific PRO-C3 ELISA measures true formation of type III collagen associated with liver and muscle parameters. Am J Transl Res. 2013 Apr 19;5(3):303-15. Print 2013. PMID 23634241
- [Background] Nielsen MJ, Veidal SS, Karsdal MA, Orsnes-Leeming DJ, Vainer B, Gardner SD, Hamatake R, Goodman ZD, Schuppan D, Patel K. Plasma Pro-C3 (N-terminal type III collagen propeptide) predicts fibrosis progression in patients with chronic hepatitis C. Liver Int. 2015 Feb;35(2):429-37. doi: 10.1111/liv.12700. Epub 2014 Oct 29. PMID 25308921
- [Background] Helmke S, Colmenero J, Everson GT. Noninvasive assessment of liver function. Curr Opin Gastroenterol. 2015 May;31(3):199-208. doi: 10.1097/MOG.0000000000000167. PMID 25714706
- [Background] Schnabl B, Brenner DA. Interactions between the intestinal microbiome and liver diseases. Gastroenterology. 2014 May;146(6):1513-24. doi: 10.1053/j.gastro.2014.01.020. Epub 2014 Jan 15. PMID 24440671
- [Background] Bonder A, Afdhal N. Utilization of FibroScan in clinical practice. Curr Gastroenterol Rep. 2014 Feb;16(2):372. doi: 10.1007/s11894-014-0372-6. PMID 24452634
- [Background] Chen J, Talwalkar JA, Yin M, Glaser KJ, Sanderson SO, Ehman RL. Early detection of nonalcoholic steatohepatitis in patients with nonalcoholic fatty liver disease by using MR elastography. Radiology. 2011 Jun;259(3):749-56. doi: 10.1148/radiol.11101942. Epub 2011 Apr 1. PMID 21460032
- [Background] Thomas MS, Newman D, Leinhard OD, Kasmai B, Greenwood R, Malcolm PN, Karlsson A, Rosander J, Borga M, Toms AP. Test-retest reliability of automated whole body and compartmental muscle volume measurements on a wide bore 3T MR system. Eur Radiol. 2014 Sep;24(9):2279-91. doi: 10.1007/s00330-014-3226-6. Epub 2014 May 29. PMID 24871333
- [Background] Karlsson A, Rosander J, Romu T, Tallberg J, Gronqvist A, Borga M, Dahlqvist Leinhard O. Automatic and quantitative assessment of regional muscle volume by multi-atlas segmentation using whole-body water-fat MRI. J Magn Reson Imaging. 2015 Jun;41(6):1558-69. doi: 10.1002/jmri.24726. Epub 2014 Aug 11. PMID 25111561
- [Background] West J, Dahlqvist Leinhard O, Romu T, Collins R, Garratt S, Bell JD, Borga M, Thomas L. Feasibility of MR-Based Body Composition Analysis in Large Scale Population Studies. PLoS One. 2016 Sep 23;11(9):e0163332. doi: 10.1371/journal.pone.0163332. eCollection 2016. PMID 27662190
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- See also: Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 7/18/2018 and concluded 12/3/2019. Participants were recruited from a local bariatric surgery medical practice.
Period: Overall Study
Arm/Group | NASH Group | Non-NASH (NAFLD or Normal) Group
Started | 4 | 10
Completed | 4 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NASH Group | Non-NASH (NAFLD or Normal) Group | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.750 (6.551) | 38.600 (9.119) | 39.21 (8.276)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 8 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Liver Fat Between Baseline and 12 Weeks Post-surgery
Description: Assessed by magnetic resonance imaging proton density fat fraction (MRI PDFF)
Time Frame: 12 weeks
Population: Only the NASH group had longitudinal evaluation
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NASH Group | Non-NASH (NAFLD or Normal) Group
Number analyzed (Participants) | 4 | 0
percent change | -16.4 (52.9) |

2. Primary Outcome: Percent Change in Liver Stiffness Between Baseline and12 Weeks Post-surgery
Description: We will evaluate change in liver stiffness, a surrogate for fibrosis, as assessed by magnetic resonance elastography (MRE)
Time Frame: 12 weeks
Population: Only NASH group had longitudinal evaluation
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NASH Group | Non-NASH (NAFLD or Normal) Group
Number analyzed (Participants) | 4 | 0
percent change | 1.9 (10.4) |

ADVERSE EVENTS:
Time Frame: 2.22 years
Arm/Group | NASH Group | Non-NASH (NAFLD or Normal) Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 2/4 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NASH Group (N=4) | Non-NASH (NAFLD or Normal) Group (N=10)
Bruising, tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cyst in pituitaty (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gas Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
H. Pylori Infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1)
Inactive mild gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Migraine (General disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right Arm Tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Urinary Tract Infections (Infections and infestations) | 0 (0) | 1 (1)
Vitamin D Defficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Worsening Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was limited by the need to close the trial prior to enrolling all participants due to extreme difficulties with recruitment. Based on our power estimates, we needed 25 people in the NASH group, and we were only able to enroll 4. Therefore, our analyses will be limited the basic plans proposed in the protocol and will likely be exploratory and hypothesis generating in nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03294850/Prot_SAP_000.pdf